CLINICAL TRIAL: NCT02529215
Title: Improving the Quality of Team Training and Performance During Interprofessional in Situ Mock Code Blue Simulations: A Randomized Controlled Mixed-methods Study
Brief Title: Improving Team Training During Mock Code Blue Simulations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Catharine Walsh, Educational Researcher, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1000048092
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Education, Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Just-in-time training (JITT) group (Experimental): Receive a 20min just-in-time simulation-based teaching session targeting: (1) CPR quality and (2) medication administration within 3 hours of the scheduled in situ simulation.
  Interventions: Behavioral: Just-in-time training (JITT)
- No additional training (control) group (No Intervention): Control group who receives no additional training.

INTERVENTIONS:
Behavioral: Just-in-time training (JITT) — The JITT training is a 20 minute simulation-based teaching session targeting: (1) CPR quality and (2) medication administration.
  Arms: Just-in-time training (JITT) group

SUMMARY:
Communication and teamwork failures are the leading causes of errors in healthcare settings. In situ mock code simulations are a potential means to train team-based skills using simulation within real clinical care environments where errors occur; however, debriefing discussions often focus on gaps in learners' clinical skills as opposed to team functioning. This study aims to determine whether learners who are pre-trained using just-in-time simulation regarding CPR quality and medication administration will exhibit improved performance with respect to these skills during in situ mock codes as well as improved team functioning.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals, including nurses, pediatric residents, physicians and/or respiratory therapists scheduled to participate in interprofessional, team-based in situ mock codes.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Team-based non-technical skills | Time Frame: All data will be collected during the one hour when participants engage in the in situ mock code simulation
  Measured using the Team Emergency Assessment Measure (TEAM) scale

SECONDARY OUTCOMES:
CPR quality | Time Frame: All data will be collected during the one hour when participants engage in the in situ mock code simulation
  Measured using the Zoll R series defibrillator (compressions per minute (cpm), depth in millimeters (mm), and compression fraction)

OTHER OUTCOMES:
Medication errors | Time Frame: All data will be collected during the one hour when participants engage in the in situ mock code simulation
Focus of debriefing | Time Frame: All data will be collected during the one hour when participants engage in the in situ mock code simulation
  Qualitative analysis of audio-recordings
Cognitive load | Time Frame: All data will be collected during the one hour when participants engage in the in situ mock code simulation
  Measured using the Paas scale, Cognitive Load Component Questionnaire, and NASA-TLX cogntiive load questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Catharine M Walsh, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children (SickKids), Toronto, Ontario, Canada